CLINICAL TRIAL: NCT06950697
Title: Development and Application of a Thrombosis Risk Prediction Model in Lung Cancer Patients Treated With Immune Checkpoint Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Capital Medical University (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Fourth Hospital of Inner Mongolia Autonomous Region (Unknown)
Responsible Party: Sponsor
Other Study IDs: CYHF202212
Record Dates: First submitted 2025-04-08; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Venous Thromboembolism; Arterial Thromboembolism
MeSH Terms: conditions — Lung Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- with immune checkpoint inhibitor-associated venous thromboembolism: patients with immune checkpoint inhibitor-associated venous thromboembolism would be included in this group
- without immune checkpoint inhibitor-associated venous thromboembolism: patients without immune checkpoint inhibitor-associated venous thromboembolism would be included in this group
- with immune checkpoint inhibitor-associated arterial thromboembolism: patients with immune checkpoint inhibitor-associated arterial thromboembolism would be included in this group
- without immune checkpoint inhibitor-associated arterial thromboembolism: patients without immune checkpoint inhibitor-associated arterial thromboembolism would be included in this group

SUMMARY:
The purpose of this observational study is to explore the incidence, risk factors, and relationship with therapeutic outcomes of VTE (venous thromboembolism) and ATE (arterial thromboembolism) associated with immune checkpoint inhibitors (ICIs) therapy. The primary questions it aims to address are:

1. What is the real-world incidence of VTE/ATE in lung cancer patients receiving immune checkpoint inhibitors?
2. What are the risk factors for VTE/ATE in lung cancer patients receiving immune checkpoint inhibitors?
3. What is the impact of VTE/ATE on the prognosis of lung cancer patients receiving immune checkpoint inhibitors?

Researchers will compare the characteristics and biomarkers of patients with and without ICI-associated VTE/ATE to identify novel specific biomarkers for thrombotic events. Furthermore, they will construct a risk assessment model for thrombotic events to provide guidance for precision prevention and treatment in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histopathologically confirmed lung cancer diagnosis at enrollment
* Received at least one dose of a China-approved lung cancer immune checkpoint inhibitor
* Signed informed consent form

Exclusion Criteria:

* Excluded based on inclusion criteria
* Cannot comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histopathologically confirmed lung cancer who were treated with immune checkpoint inhibitors between January 1, 2019, and December 31, 2026.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune checkpoint inhibitor-associated venous thromboembolism/arterial thromboembolism | From the date of the administration of the first dose of immune checkpoint inhibitors until three months after the completion of therapy or the initiation of other anti-tumor therapies, whichever comes first, assessed up to 96 months.
  From the administration of the first dose of immune checkpoint inhibitors until three months after the completion of immune checkpoint inhibitor therapy, or until the initiation of other anti-tumor therapies following immune checkpoint inhibitor therapy, symptomatic and incidentally detected arterial thromboembolism and venous thromboembolism events that occur during this period are included.

SECONDARY OUTCOMES:
Progression-free survival | From the date of the administration of the first dose of immune checkpoint inhibitors until the date of disease progression, death from any cause, or the cutoff date, whichever comes first, assessed up to 96 months.
  Progression-Free Survival refers to the time from the start of immune checkpoint inhibitor therapy until the disease progresses or the patient dies, whichever occurs first.
Overall survival | From the date of the administration of the first dose of immune checkpoint inhibitors until the date of death from any cause, or the cutoff date, whichever comes first, assessed up to 96 months.
  Overall survival refers to the time from the start of immune checkpoint inhibitor therapy until the patient dies or the cutoff date, whichever occurs first."
Objective response rate | From the date of the first dose of immune checkpoint inhibitors until the best efficacy is achieved, assessed up to 96 months.
  Objective Response Rate (ORR) refers to the proportion of patients who experience a confirmed reduction in tumor size or complete disappearance of the tumor, as assessed by standard criteria such as RECIST (Response Evaluation Criteria in Solid Tumors). It includes both complete responses (CR) and partial responses (PR) and is typically reported as a percentage of the total treated population.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Fourth Hospital of Inner Mongolia Autonomous Region, Hohhot, Inner Mongolia
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - China-japan Friendship Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No